CLINICAL TRIAL: NCT03946917
Title: A Multi-center, Open-label, Phase I/II Clinical Trial of Tolerability, Safety and Efficacy of Recombinant Humanized Anti-PD-1 Monoclonal Antibody for Injection (JS001) Combined With Regorafenib in Patients With Advanced Colorectal Cancer
Brief Title: JS001 Combined With Regorafenib in Patients With Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Principal Investigator, Ruihua Xu, Professor, Principal Investigator, President, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS001/Regorafenib in mCRC
Record Dates: First submitted 2019-04-14; First posted 2019-05-13 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Colorectal Cancer
Keywords: Regorafenib; JS001; Colorectal cancer; Microsatellite stability
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Injections; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JS001/regorafenib (Experimental): recombinant humanized anti-PD-1 monoclonal antibody for injection (JS001) in combination with regorafenib tablet
  Interventions: Drug: JS001; Drug: regorafenib tablet

INTERVENTIONS:
Drug: JS001 — JS001 3 mg/kg, iv drip, d1, d15, q4w
  Other Names: recombinant humanized anti-PD-1 monoclonal antibody for injection
Drug: regorafenib tablet — 80/120/160 mg, po, d1-d21, Q4w.
  Other Names: STIVARGA

SUMMARY:
Colorectal cancer is one of the most common malignancies in China. Regorafenib is the standard multi-kinase inhibitor for refractory advanced colorectal cancer. In mice, regorafenib combined with anti-PD-1 was shown superior to regorafenib, which has not yet been verified in humans. JS001 is the Chinese anti-PD-1 monoclonal antibody for injection which has been approved for melanoma. This study is the first multi-center, open-label, phase I/II clinical trial to evaluate tolerability, safety and efficacy of JS001 in combination with regorafenib tablet in patients with MSS/MSI-L/pMMR, relapsed or metastatic colorectal cancer who have failed or can not tolerate fluorouracil, oxaliplatin and irinotecan based systemic treatment. The phase I clinical trial is to determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of regorafenib tablet in this regimen, and select an acceptable safe dose for the phase II clinical trial to further determine safety and efficacy of this combination regimen in patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
Colorectal cancer is one of the most common malignancies in China, with incidence and mortality ranking the 3rd and 4th among malignancies in China. Regorafenib is the standard multi-kinase inhibitor for refractory metastatic colorectal cancer, with multiple anti-tumor effects by inhibiting targets related to tumor cell proliferation, tumor metastasis, tumor angiogenesis and tumor immune escape, howerver, its efficacy is limited. Immunotherapy has become standard treatment for mCRC patients with MSI-H/dMMR. Combination of anti-angiogenesis treatment and immunotherapy may have a better anti-tumor effect. In mice, regorafenib combined with anti-PD-1 was shown superior to regorafenib, which has not yet been verified in humans. JS001 is the Chinese anti-PD-1 monoclonal antibody for injection which has been approved for melanoma. This study is the first multi-center, open-label, phase I/II clinical trial to evaluate tolerability, safety and efficacy of JS001 in combination with regorafenib tablet in patients with MSS/MSI-L/pMMR, relapsed or metastatic colorectal cancer who have failed or can not tolerate fluorouracil, oxaliplatin and irinotecan based systemic treatment. The phase I clinical trial is to determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of regorafenib tablet in this regimen, and select an acceptable safe dose for the phase II clinical trial to further determine safety and efficacy of this combination regimen in patients with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged ≥18 years;
2. Histologically or cytologically confirmed colon or rectal adenocarcinoma, with unresectable relapsed or metastatic disease;
3. Microsatellite stability (MSS) or microsatellite instability-low (MSI-L), or proficient expression of DNA mismatch repair gene (pMMR);
4. Patients who have failed, or can not tolerate after previous systemic treatment for relapsed or metastatic colorectal cancer, with no more than 3 months for disease progression after the last systemic treatment. The systemic treatment must contain fluorouracil, oxaliplatin and irinotecan, with or without targeted therapy (bevacizumab, cetuximab, and so on);
5. With at least 1 measurable lesion according to RECIST 1.1 criteria; 1) Non-nodal lesions with the maximum diameter ≥10mm, or nodal lesions with the short axis ≥15mm; 2) For lesions previously treated locally with radiotherapy or ablation, if there is definite progression according to RECIST 1.1, and the maximum diameter ≥10mm, these can also be considered as measurable target lesions.
6. ECOG score 0-1;
7. Expected survival ≥3 months;
8. Good organ function (without blood transfusion, use of hematopoietic stimulating factors, or transfusion of albumin or blood products within 14 days prior to examination):

1) Platelet (PLT) count ≥100,000 /mm3; 2) Neutrophil count (ANC) ≥1,500 /mm3; 3) Hemoglobin (Hb) level ≥9.0 g/dl; 4) International normalized ratio (INR) ≤1.5; 5) Prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤1.5×ULN; 6) Glycosylated hemoglobin (HbA1c) <7.5%; 7) Total bilirubin (TBIL) level ≤1.5×ULN; 8) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) level ≤2.5×ULN (≤5×ULN in case of liver metastasis); 9) Alkaline phosphatase level ≤2.5×ULN (≤5×ULN in case of liver metastasis); 10) Serum creatinine (Cr) level ≤1.5×ULN and creatinine clearance ≥60 ml/min; 11) Thyroid stimulating hormone (TSH) ≤ULN; 12) Normal serum free thyroid hormone (T4); 13) Normal serum free triiodothyronine (T3); 14) Serum amylase ≤1.5×ULN; 15) Lipase ≤1.5×ULN. 9. Females of child bearing age must have a negative pregnancy test, and have to take contraception measures and avoid breast feeding during the study and for 3 months after the last dose; male subjects must agree to taken contraception measures during the study and for 3 months after the last dose.

10. Able to understand and willing to sign written informed consent form.

Exclusion Criteria:

1. Diagnosis of any other malignancy at different primary site or of different histological type from colorectal cancer within 5 years prior to initiation of study treatment, except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of cervix;
2. Microsatellite instability-high (MSI-H) or deficient expression of DNA mismatch repair gene (dMMR);
3. Previous treatment with regorafenib, PD-1/PD-L1/PD-L2 antibody or any other antibody that acts on T cell costimulatory or checkpoint pathways;
4. Known allergy to study drug or excipients, or allergy to similar drugs;
5. Have received other anti-tumor treatment within 4 weeks prior to initiation of study treatment, or no more than 5 half lives from the last dose;
6. Have participated in other clinical study and received drug within 4 weeks prior to initiation of study treatment;
7. Have undergone major surgery or open biopsy, or have massive trauma within 4 weeks prior to initiation of study treatment;
8. Have received immunosuppressants (excluding inhaled corticosteroids or ≤10 mg/day prednisone or other systemic steroids at equivalent pharmaphysiological dose) within 2 weeks prior to initiation of study treatment;
9. Have vaccination with attenuated live vaccines within 4 weeks prior to initiation of the study treatment or plan to vaccinate during the study;
10. CYP3A4 inducers or inhibitors should not be stopped within 1 week prior to initiation of study treatment and during the study;
11. Known metastasis to central nervous system;
12. Present or history of any autoimmune disease;
13. Human immunodeficiency virus (HIV) infection (HIV antibody positive), or active hepatitis C virus (HCV) infection (HCV antibody positive), or active hepatitis B virus (HBV) infection (HBsAg or HBcAb positive, and HBV-DNA ≥2000 IU/ml (copies/ml)), or other severe infection requiring systemic antibiotic treatment, or unexplained body temperature >38.5℃ during screening period/before study treatment;
14. Presence of pleural effusion, peritoneal effusion, or pericardial effusion;
15. Development of the following diseases within 6 months prior to initiation of study treatment: myocardial infarction, severe/unstable angina, congestive heart failure above NYHA grade 2, poorly controlled arrhythmia;
16. Poorly controlled hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg);
17. With bleeding tendency, or evident hemoptysis or other hemorrhagic events (e.g. gastrointestinal hemorrhage, hemorrhagic gastric ulcer) within 2 months prior to initiation of study treatment, or presence of hereditary or acquired bleeding or thrombotic tendency (e.g. hemophilia, coagulopathy, thrombocytopenia, etc.), or current/long-term thrombolytic or anticoagulant therapy (except aspirin ≤100 mg/day);
18. Development of arterial/venous thrombotic events, e.g. cerebrovascular accident (transient ischemic attack, cerebral hemorrhage, cerebral infarction etc.), deep venous thrombosis, vasculitis, etc. within 6 months prior to initiation of study treatment;
19. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
20. Seizure requiring drug (e.g. steroids or antiepileptic drugs) treatment;
21. Presence of malabsorption disorder;
22. Unable to swallow study drug;
23. Presence of toxicities (except alopecia) of grade 2 and above (CTCAE V5.0) due to previous anti-tumor treatment or surgical procedure;
24. History of drug abuse, illegal drug use or alcohol dependence;
25. Patients with other severe acute or chronic conditions that may increase the risk of participation in the study and study treatment, or may interfere with interpretation of study results, and judged by the investigator as not suitable for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2021-11-20 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 28 days after the first dose of JS001 and Regorafenib, assessed up to 8 months
  The maximum dose that patients enrolled can tolerate during dose escalation of phase I clinical trial according to mTPI method
Dose limiting toxicity (DLT) | 28 days after the first dose of JS001 and Regorafenib, assessed up to 8 months
  Severe toxicity that may be related to JS001 or regorafenib during dose escalation of phase I clinical trial according to mTPI method
Objective response rate (ORR) | from the initiation date of first cycle to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  The ratio of patients who are evaluated as CR or PR

SECONDARY OUTCOMES:
Progression free survival (PFS) | from the initiation date of first cycle to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  The Kaplan-Meier survival from the initiation date of first cycle until the date of first documented progression or date of death
Overall survival (OS) | from the initiation date of first cycle to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  The Kaplan-Meier survival from the initiation date of first cycle until death from any cause or the last follow-up date.
Disease control rate (DCR) | from the initiation date of first cycle to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Defined as the proportion of patients whose tumors shrink or remain stable for a certain period of time, including CR, PR and SD.
Duration of response (DOR) | the first assessment of a tumor as PR or CR and the first assessment as PD or any cause of death or the last follow-up date, assessed up to 2 years.
  defined as the time between the first assessment of a tumor as PR or CR and the first assessment as PD or any cause of death
Severe toxicity | from the initiation date of first cycle to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  ≥ Grade 3 toxicities
cfDNA | from the initiation date of first cycle to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  The dynamic variation of circulating free DNA or cell free DNA (cfDNA) in immunotherapy efficacy and safety assessment
Intestinal microorganism | from the initiation date of first cycle to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  The composition of intestinal microorganism pre- and post-treatment tested by intestinal microorganism, the relationship between intestinal flora alpha diversity and beta diversity and immunotherapy response as well as between intestinal microorganism alpha diversity and beta diversity and treatment toxicity and tolerance.

CONTACTS AND LOCATIONS:
Overall Officials: Rui-hua Xu, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yoshino T, Komatsu Y, Yamada Y, Yamazaki K, Tsuji A, Ura T, Grothey A, Van Cutsem E, Wagner A, Cihon F, Hamada Y, Ohtsu A. Randomized phase III trial of regorafenib in metastatic colorectal cancer: analysis of the CORRECT Japanese and non-Japanese subpopulations. Invest New Drugs. 2015 Jun;33(3):740-50. doi: 10.1007/s10637-014-0154-x. Epub 2014 Sep 12. PMID 25213161
- [Result] Li J, Qin S, Xu R, Yau TC, Ma B, Pan H, Xu J, Bai Y, Chi Y, Wang L, Yeh KH, Bi F, Cheng Y, Le AT, Lin JK, Liu T, Ma D, Kappeler C, Kalmus J, Kim TW; CONCUR Investigators. Regorafenib plus best supportive care versus placebo plus best supportive care in Asian patients with previously treated metastatic colorectal cancer (CONCUR): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2015 Jun;16(6):619-29. doi: 10.1016/S1470-2045(15)70156-7. Epub 2015 May 13. PMID 25981818
- [Result] McDermott DF, Sosman JA, Sznol M, Massard C, Gordon MS, Hamid O, Powderly JD, Infante JR, Fasso M, Wang YV, Zou W, Hegde PS, Fine GD, Powles T. Atezolizumab, an Anti-Programmed Death-Ligand 1 Antibody, in Metastatic Renal Cell Carcinoma: Long-Term Safety, Clinical Activity, and Immune Correlates From a Phase Ia Study. J Clin Oncol. 2016 Mar 10;34(8):833-42. doi: 10.1200/JCO.2015.63.7421. Epub 2016 Jan 11. PMID 26755520
- [Result] Tang B, Yan X, Sheng X, Si L, Cui C, Kong Y, Mao L, Lian B, Bai X, Wang X, Li S, Zhou L, Yu J, Dai J, Wang K, Hu J, Dong L, Song H, Wu H, Feng H, Yao S, Chi Z, Guo J. Safety and clinical activity with an anti-PD-1 antibody JS001 in advanced melanoma or urologic cancer patients. J Hematol Oncol. 2019 Jan 14;12(1):7. doi: 10.1186/s13045-018-0693-2. PMID 30642373
- [Result] Yaghoubi N, Soltani A, Ghazvini K, Hassanian SM, Hashemy SI. PD-1/ PD-L1 blockade as a novel treatment for colorectal cancer. Biomed Pharmacother. 2019 Feb;110:312-318. doi: 10.1016/j.biopha.2018.11.105. Epub 2018 Dec 3. PMID 30522017